CLINICAL TRIAL: NCT01074840
Title: Dendritic Cell Responses to Viral Stimulation in Peanut Allergic Subjects Undergoing Peanut Oral Immunotherapy
Brief Title: Understanding How the Immune System Responds to Viruses in Peanut Allergic Children Undergoing Peanut Oral Immunotherapy
Acronym: DCOIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Drew Bird, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112009-006
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Peanut Allergy
Keywords: Food Hypersensitivity; Hypersensitivity; Immune System Diseases; Hypersensitivity, Immediate; Peanut Hypersensitivity; Food Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity; Immune System Diseases; Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut (Active Comparator): Peanut flour will be given in increasing amounts.
  Interventions: Other: Peanut flour
- Control (No Intervention): Subjects will be enrolled who meet the inclusion/exclusion criteria and followed as matched controls. These subjects will not receive any treatment.

INTERVENTIONS:
Other: Peanut flour — Peanut-allergic subjects will be given peanut flour in increasing amounts.
  Arms: Peanut

SUMMARY:
The purpose of this study is to find out if there is a way to treat children with peanut allergy to help lower the risk of severe allergic reactions and also cause them to lose their allergy to peanuts and to understand what happens to their immune systems when they have viral infections while on therapy. The approach we will use to treat peanut allergy in this study is a process called desensitization.

We think that children with a peanut allergy receiving peanut oral immunotherapy will be able to eat more peanuts without having a reaction by the end of the study than they could eat at the beginning. We also think that we will be able to measure changes in their immune system and their immune system's response to viruses while they are on therapy.

DETAILED DESCRIPTION:
Peanut allergy is known to cause severe anaphylactic reactions. Compared with other food allergies it tends to be more persistent and also its prevalence seems to be rising. Currently there is no proven treatment other than strict avoidance. We are attempting to decrease the risk of anaphylaxis on accidental ingestion by desensitizing subjects to peanut using peanut oral immunotherapy (OIT). We are also studying the effect of viral infections on the immune system in children receiving peanut OIT.

Children ages three to sixteen years of age with peanut allergy will be given peanut OIT. Twenty-five subjects will also be recruited as controls. These subjects will not receive any peanut or placebo but only have skin prick testing and lab work in addition to a history and physical exam. Active subjects will undergo a double-blind food challenge at entry to verify that they are allergic to peanuts. If allergic, they will then have modified rush immunotherapy on the first day and then increase the doses at least every two weeks up to a maintenance dose of 4 grams (equivalent to about 13 peanuts). Doses will be taken daily at home except for dose increases which will be done at Children's Medical Center. Outcome variables of interest include response to double-blind placebo controlled food challenge, skin prick testing, peanut specific IgE, and adverse events. These results will be compared between the start and end of peanut OIT using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 16 years of either sex, any race, any ethnicity, weighing at least 18.3 kg at the time of the initial visit.
* The presence of IgE specific to peanuts (a positive skin prick test to peanuts (diameter of wheal > 3.0 mm) and a positive in vitro IgE (CAP-FEIA) > 7 kU/L) measured within the past year.
* Significant clinical symptoms occurring within 60 minutes after ingesting peanuts during an observed Double-Blind Placebo Controlled Food Challenge.
* Provide signed informed consent.
* Ability to follow-up regularly for scheduled appointments.
* Females of child-bearing potential must be willing to practice an acceptable form of birth control throughout the protocol.

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise (Cyanosis or SpO2 < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence)
* Currently participating in a study using an investigational new drug.
* Participation in any interventional study for the treatment of food allergy in the past 12 months or while participating in this study.
* Subjects with a known oat or wheat (because of potential cross contamination with oat) food allergy will be excluded
* Poor control or persistent activation of atopic dermatitis.
* Diagnosis of asthma and currently being treated with daily doses of inhaled corticosteroids or requiring a rescue inhaler more than 2 days per week.
* Inability to discontinue antihistamines for skin testing and Oral Food Challenges (OFCs).
* Pregnant female.
* Chronic medical condition requiring frequent use of oral steroids, chronic psychiatric illness or history of substance abuse.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
We will measure changes in the immune system on a molecular level affected by viral infections in peanut allergic children undergoing peanut OIT. | 5 years

SECONDARY OUTCOMES:
We will determine if our peanut OIT protocol lowers the risk of anaphylaxis in peanut allergic children. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John A Bird, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center Dallas Food Allergy Center, Dallas, Texas, United States

REFERENCES:
- [Result] Jones SM, Pons L, Roberts JL, Scurlock AM, Perry TT, Kulis M, Shreffler WG, Steele P, Henry KA, Adair M, Francis JM, Durham S, Vickery BP, Zhong X, Burks AW. Clinical efficacy and immune regulation with peanut oral immunotherapy. J Allergy Clin Immunol. 2009 Aug;124(2):292-300, 300.e1-97. doi: 10.1016/j.jaci.2009.05.022. Epub 2009 Jul 3. PMID 19577283
- [Result] Hofmann AM, Scurlock AM, Jones SM, Palmer KP, Lokhnygina Y, Steele PH, Kamilaris J, Burks AW. Safety of a peanut oral immunotherapy protocol in children with peanut allergy. J Allergy Clin Immunol. 2009 Aug;124(2):286-91, 291.e1-6. doi: 10.1016/j.jaci.2009.03.045. Epub 2009 May 27. PMID 19477496